CLINICAL TRIAL: NCT02568059
Title: The Clinical Safety of Alcoholic Extract Sahastara Remedy of Extract Capsule in Healthy Volunteers (Clinical Trial Phase I)
Brief Title: The Clinical Safety of Alcoholic Extract Sahastara Remedy of Extract Capsule in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Thammasat University (Other)
Responsible Party: Principal Investigator, Puritat Kanokkangsadal, Department of Applied Thai Traditional Medicine, Faculty of Medicine, Thammasat University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MTU-EC-TM-1-179/57; TCTR20150917001 (Registry Identifier: Thai Clinical Trials Registry(TCTR))
Record Dates: First submitted 2015-09-30; First posted 2015-10-05 (Estimated); Last update posted 2016-10-18 (Estimated); Status verified 2016-10

CONDITIONS: Osteoarthritis
MeSH Terms: conditions — Osteoarthritis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 100 mg SHT extract (Experimental): The Sahastara remedy alcoholic extract capsule dose 100 mg.
  Interventions: Drug: Sahastara remedy alcoholic extract
- 200 mg SHT extract (Experimental): The Sahastara remedy alcoholic extract capsule dose 200 mg.
  Interventions: Drug: Sahastara remedy alcoholic extract

INTERVENTIONS:
Drug: Sahastara remedy alcoholic extract — comparison of different dose of drug

SUMMARY:
The clinical safety of Sahastara remedy alcoholic extract in healthy volunteers. Investigators will investigate safety of 100 and 200 mg of Sahastara remedy extract capsule in healthy volunteers. This is Clinical trial Phase I.

DETAILED DESCRIPTION:
The sahastara remedy (SHT) is a Thai traditional medicine that is use to relieve pain of musculoskeletal problem. There is study shown that SHT extract was not found acute and chronic toxicity in rat. However, there is no study regarding safety in human. Thus, this study is a clinical trial Phase I that investigate clinical safety of SHT alcoholic extract in healthy volunteers. The clinical safety will monitor for 28 days in continuously use of 100 and 200 mg SHT extraction 3 time a day and after stop intervention for 14 days.

ELIGIBILITY:
Inclusion Criteria:

* No pregnancy
* No Serious Medical Condition evaluated by Physical Examination and Laboratory results in 1 month before study
* No Supplementary food and/or Vitamin during the study
* Able to follow suggestion during the study

Exclusion Criteria:

* Uncontrolled Hypertension (BP>140/90 mm.Hg.)
* BMI > 30
* Have serious medical condition including Severe peptic ulcer, congestive heart disease, Liver and Renal dysfunction.
* On during use medicine including Rifampicin, Phenytoin, Propranolol, Theophylline

Ages: 20 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 25 (Actual)
Dates: Start 2015-12; Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Clinical safety evaluated by History taking, Patient diary note, Physical Examination and Laboratory test including Complete Blood Count (CBC), Renal functions, Liver functions, Lipid profile, Fasting Blood Sugar (FBS), and Urinary analysis | 14 days while using intervention
  Clinical safety was evaluated changing from baseline by History taking, Patient diary note, Physical Examination and Laboratory test including Complete Blood Count (CBC), Renal functions, Liver functions, Lipid profile, Fasting Blood Sugar (FBS), and Urinary analysis
Clinical safety evaluated by History taking, Patient diary note, Physical Examination and Laboratory test including Complete Blood Count (CBC), Renal functions, Liver functions, Lipid profile, Fasting Blood Sugar (FBS), and Urinary analysis | 28 days while using intervention
  Clinical safety was evaluated changing from baseline and 14 days while using intervention by History taking, Patient diary note, Physical Examination and Laboratory test including Complete Blood Count (CBC), Renal functions, Liver functions, Lipid profile, Fasting Blood Sugar (FBS), and Urinary analysis
Clinical safety evaluated by History taking, Patient diary note, Physical Examination and Laboratory test including Complete Blood Count (CBC), Renal functions, Liver functions, Lipid profile, Fasting Blood Sugar (FBS), and Urinary analysis | 14 days after stop intervention
  Clinical safety was evaluated changing from baseline,14 days and 28 days while using intervention by History taking, Patient diary note, Physical Examination and Laboratory test including Complete Blood Count (CBC), Renal functions, Liver functions, Lipid profile, Fasting Blood Sugar (FBS), and Urinary analysis

CONTACTS AND LOCATIONS:
Overall Officials: Puritat Kanokkangsadal, M.Sc., Principal Investigator — Department of Applied Thai Traditional Medicine, Faculty of Medicine, Thammasat University
Locations (1):
- Faculty of Medicine, Thammasat University, Klongnueng, Changwat Pathum Thani, Thailand